CLINICAL TRIAL: NCT03196882
Title: Effectiveness of Adaptation of the Dose of Iron Supplementation in Pregnancy on Maternal-child Health. Randomized Clinical Trial (ECLIPSES)
Brief Title: Effectiveness of Adaptation of the Dose of Iron Supplementation in Pregnancy on Maternal-child Health. (ECLIPSES)
Acronym: (ECLIPSES)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Victoria Arija Val (Other)
Collaborators: University Rovira i Virgili (Other); Catalan Institute of Health (Other Government); Hospital Universitari Joan XXIII de Tarragona. (Other); Carlos III Health Institute (Other Government)
Responsible Party: Sponsor-Investigator, Victoria Arija Val, Professor, MD, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Organization: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IJG-FER-2012; 2012-005480-28 (EudraCT Number); PI12/02777 (Other Grant/Funding Number: Instituto de Salud Carlos III,Ministerio de Sanidad)
Record Dates: First submitted 2017-06-15; First posted 2017-06-23 (Actual); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Anemia Ferropenic; Risk of Hemoconcentration (Iron Levels >130g/L)
Keywords: pregnancy; iron; hemoglobin; supplementation; neurodevelopment; newborn; anemia; clinical trial
MeSH Terms: conditions — Anemia | interventions — Iron

STUDY DESIGN:
Intervention Model Description: Multi-centered, parallel groups, controlled, triple blind, randomized clinical trial (RCT) subdivided in 2 strata as a function of the hemoglobin (Hb) levels at the start of the pregnancy:
  Stratum 1: If Hb from 110 to 130 g/L, randomly assigned at week 12 to receive iron supplement of 40 or 80 mg/d.
  Stratum 2: If Hb >130 g/L, randomly assigned at week 12 to receive iron supplement of 40 or 20 mg/d.
  The study is structured as a RCT with 2 stratum, depending on the Hb levels before week 12 of gestation. In each stratum there are two arms of intervention. Total 4 arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be triple blind: the participant, the health-care professional, and the investigator-statistician. The treatment drug will be administered "blind" i.e. the doses are not identifiable since the packaging has the same format, presentation, and visual characteristics. For Stratum 1, the treatments will be designated as A or B, and for Stratum 2 they will be designated as C or D. The laboratory of MEIJI TEDEC FARMA, SA will be responsible for manufacturing, packaging and labeling the study medications. Only MEIJI TEDEC FARMA, SA and the Clinical Pharmacology Service of the Vall d'Hebron Hospital in Barcelona will know the distribution codes and the composition of each of the treatments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stratum 1: 40 mg/day of iron (Active Comparator): Ferrimanitol ovoalbumin. 40mg of iron in a sachet (powder for oral solution) by mouth, every 24 hours from 12th week of gestation to partum
  Stratum 1: If the levels of Hb are situated between 110 and 130 g/L, the individual will be randomly assigned to an iron dose supplement of 40 (medium supplementation) or 80 mg/d (high supplementation)
  Interventions: Drug: 40mg/day of iron
- Stratum 1: 80 mg/day of iron (Experimental): Ferrimanitol ovoalbumin. 80mg of iron in a sachet (powder for oral solution) by mouth, every 24 hours from 12th week of gestation to partum
  Stratum 1: If the levels of Hb are situated between 110 and 130 g/L, the individual will be randomly assigned to an iron dose supplement of 40 (medium supplementation) or 80 mg/d (high supplementation)
  Interventions: Drug: 80mg/day of iron
- stratum 2: 40 mg/day of iron (Active Comparator): Ferrimanitol ovoalbumin. 40mg of iron in a sachet (powder for oral solution) by mouth, every 24 hours from 12th week of gestation to partum
  Stratum 2: If the levels of Hb are >130 g/L, the individual will be randomly assigned to an iron dose supplement of 40 (medium supplementation) or 20 mg/d (low supplementation)
  Interventions: Drug: 40mg/day of iron
- stratum 2: 20 mg/day of iron (Experimental): Ferrimanitol ovoalbumin. 20mg of iron in a sachet (oral solution) by mouth, every 24 hours from 12th week of gestation to partum
  Stratum 2: If the levels of Hb are >130 g/L, the individual will be randomly assigned to an iron dose supplement of 40 (medium supplementation) or 20 mg/d (low supplementation)
  Interventions: Drug: 20mg/day of iron

INTERVENTIONS:
Drug: 40mg/day of iron — Ferrimanitol ovalbumin granulated. Powder for oral solution. The doses of 40 mg per day of elemental iron correspond to 300 mg ferrimanitol ovoalbumin
  Other Names: PROFER 40 mg
  Arms: Stratum 1: 40 mg/day of iron; stratum 2: 40 mg/day of iron
Drug: 20mg/day of iron — Ferrimanitol ovalbumin granulated Powder for oral solution. The doses of 20 mg per day of elemental iron correspond to 150 mg ferrimanitol ovoalbumin
  Other Names: FERROPROTINA
  Arms: stratum 2: 20 mg/day of iron
Drug: 80mg/day of iron — Ferrimanitol ovalbumin granulated. Powder for oral solution The doses of 80 mg per day of elemental iron correspond to 600 mg ferrimanitol ovoalbumin.
  Other Names: PROFER 80 mg
  Arms: Stratum 1: 80 mg/day of iron

SUMMARY:
Currently, there is no consensus regarding iron supplementation dose that is most beneficial for maternal and offspring health during gestation. This deficit, or excess, of iron prejudices the mother-child wellbeing. Therefore the hypotheses are that an iron supplementation adapted to values of hemoglobin at the start of the pregnancy will would be more effective in preventing iron deficiency, without increasing the risk of hemoconcentration by the end of pregnancy. This would be helped optimize mother-child health status.

The aims of the study are to determine the highest level of effectiveness of iron supplementation adapted to hemoglobin (Hb) levels in early pregnancy, which would be optimum for mother-child health.

To accomplish this objective a Randomized Clinical Trial (RCT) triple-blinded was designed. The study is structured as a RCT with 2 strata, depending on the Hb levels before week 12 of gestation.

Stratum 1: If Hb from 110 to 130 g/L, randomly assigned at week 12 to receive iron supplement of 40 or 80 mg/d.

Stratum 2: If Hb >130 g/L, randomly assigned at week 12 to receive iron supplement of 40 or 20 mg/d.

This study will be conducted in non-anemic pregnant women at early gestation stage, and their subsequent newborns. The data recollected to mothers will be: socio-economic data, clinical history, food item frequency, lifestyle and emotional state, and adherence to iron supplement prescription. In addition, biochemical measured will be Hemoglobin, serum ferritin, C reactive protein, cortisol, and alterations in the HFE gene (C282Y, H63D). In children, the data collected will be: ultrasound fetal biometry, anthropometric measurements, and temperament development

Should conclusive outcomes be reached, the study would indicate the optimal iron supplementation dose required to promote maternal and infant health. These results would contribute towards developing guidelines for good clinical practice.

DETAILED DESCRIPTION:
The study will be conducted in 2 Primary Care Centers (PCC) from Tarragona and Reus of the Catalunya Sexual and Reproductive Healthcare Service [Atención a la Salud Sexual y Reproductiva (ASSIR)] of the Catalan Institute of Health [Instituto Catalán de la Salud (ICS)]. The specialist health-care workers include gynecologists and midwives. The participating reproductive health-care services (RHS) provide cover for urban, suburban, and rural PCCs.

The clinical follow-up of the pregnancy in the PCC will be according to the program set by RHS. This includes a clinical visit at recruitment into the present study, a visit every trimester, and one at 40 days post-partum.

In the recruitment visit before week 12 of the pregnancy, the inclusion criteria will be assessed (except the Hb levels and the number of fetuses) as well as the exclusion criteria. Informed consent will be solicited. A clinical history will be recorded, which include date of birth, socioeconomic status, parity, date of last menstruation, corrected date of last menstruation, estimated date of partum, risk factors during pregnancy, pregnancy planning, previous use of contraceptives, clinical antecedents, surgery and personal obstetric data, toxic habits, blood pressure, height, weight of the mother (self-reported at the recruitment visit and measured objectively at each clinical follow-up visit). Similar data from the father will be solicited.

Moreover, a questionnaire regarding the ingestion of iron supplements, multi-vitamins, or other treatments and, if a smoker, the Fagerstrom test for tobacco dependency. A blood sample for standard biochemical analyses (including hemoglobin) will be sent for processing in the centralized laboratory.

At visit 1, around the 12th week of gestation, Hb levels will be evaluated as will be the number of fetuses (using echography) to confirm that the inclusion criteria are fulfilled. If fulfilled, the individuals will be retained in the study and, if not, will be transferred out of the study, and considered a screening failure. The remaining women will be assigned to Stratum 1 or Stratum 2 of the study and will be randomized with respect to iron supplement prescription. Clinical history will be taken, including the use of multi-vitamins and iron supplements and the questionnaires filled-in about food consumption, physical activity, anxiety status and tobacco dependency. ). A physical examination will be performed to measure weight and blood pressure. The ultrasound data on the fetus will be recorded to assess Crown Rump Length (CRL). A physical examination will be performed to measure weight and blood pressure. Venous blood will be taken for analyses, the results of which will be reviewed in the next clinical visit. The iron supplementation that will be needed at the next visit will be prepared for distribution. Adverse events occurring since the previous visit will be recorded.

At visit 2, around week 24 of gestation, clinical history will be taken, and will include questionnaire about use of multi-vitamins and iron supplements which, from this visit onwards, includes the adherence to the iron supplementation prescribed. The questionnaires about food consumption, physical activity, anxiety status and tobacco dependency are filled-in. A physical examination will be performed to measure weight and blood pressure. The fetal ultrasound data will be registered to assess status of fetus and estimated fetal weight. The biochemical analyses/results will be reviewed and a further blood sample taken for analysis, the results of which will be reviewed at the next clinical visit. The iron supplementation that will be needed at the next visit will be prepared for distribution. Adverse events occurring since the previous visit will be recorded.

At visit 3, around week 36 of gestation, the clinical history will be taken, the questionnaire about use of multi-vitamins and iron supplements as well as the questionnaires about food consumption, physical activity, anxiety status and tobacco dependency will be filled-in. A physical examination will be performed to measure weight and blood pressure. The fetal ultrasound data will be recorded to assess status of fetus and estimated fetal weight and the biochemical results will be evaluated. A further blood sample will be taken for analyses, the results of which will be discussed at the next clinical visit. The iron supplementation that will be needed at the next visit will be prepared for distribution. Adverse events occurring since the previous visit will be recorded.

At visit 4 (40 days post-partum), the clinical history will be taken, the questionnaire about use of multi-vitamins and iron supplements as well as the questionnaires about food consumption, physical activity, anxiety status and tobacco dependency will be filled-in. A questionnaire on post-partum depression and the Parenting Stress Index will be applied. The standard laboratory analyses results will be discussed. A further blood sample will be taken for analyses. Data on birth (type of delivery) and the newborn will be recorded (weight and height). Clinical history of the baby will be recorded, including: gender, status of newborn, Apgar score, anthropometric data (weight, height, head circumference), breastfeeding and levels of vitamin D. Cognitive development will be assessed, as well as behavioral and temperament. Adverse events occurring since the previous visit will be recorded.

Sample size:

To achieve the study's main objective, sample size is calculated in accordance with the following parameters: an alpha risk of 0.05 and a beta risk of 0.20 in a two tailed test of comparison. A drop-out rate or lack of data of 35% is factored-in.

To calculate the sample size, previous data from the research group of investigators were consulted (Aranda, 2011, Hernández-Martínez, 2011, Ribot, 2012). A prevalence of 23.5% of iron deficiency anemia was observed in the 3rd trimester in pregnant women with Hb levels of 110-130 g/L in the first trimester and a prevalence of risk of hemoconcentration of 14.7% in the 3rd trimester of pregnant women who started pregnancy with Hb levels of 130-150 g/L.

* In Stratum 1, to reduce the frequency of anemia ferropenic from 23.5% to 11.5% in the intervention group supplemented with 80mg/day of iron with respect to the group supplemented with 40mg/day, will be necessary to include 236 women in each group
* In Stratum 2, to reduce the frequency of hemocontration from 14.7% to 2.7% in the intervention group supplemented with 20mg/day of iron with respect to the group supplemented with 40mg/day, will be necessary to include 116 women in each group

Intervention assignment: Allocation

The pregnant women are assigned to Stratum 1 or Stratum 2 as a function of the hemoglobin values in the baseline analysis of the study. They are, then, randomly assigned to 2 treatment groups to receive different iron supplements.

Stratum 1: If Hb from 110 to 130 g/L, randomly assigned at week 12 to receive iron supplement of 40 or 80 mg/d.

Stratum 2: If Hb >130 g/L, randomly assigned at week 12 to receive iron supplement of 40 or 20 mg/d.

The randomization is performed using centralized computer software, which is automatic and masked and applies to the electronic data collection forms, as well. The procedure for randomization is independent for each Stratum.

Blinding The study will be triple blind: the participant, the health-care professional, and the statistician. The treatment drug will be administered "blind" i.e. the doses are not identifiable since the packaging has the same format, presentation, and visual characteristics. The laboratory of MEIJI TEDEC FARMA, SA will be responsible for manufacturing, packaging and labeling the study medications.

Only MEIJI TEDEC FARMA, SA and the Clinical Pharmacology Service of the Vall d'Hebron Hospital in Barcelona will know the distribution codes and the composition of each of the treatments.

There would be no need for un-blinding except if an unexpected serious adverse event occurs. In which case, the pharmaco-vigilance staff of TEDEC-MEIJI FARMA S.A. will take responsibility for un-blinding and communicating the adverse event to the appropriate health authorities. TEDEC-Meiji Farma SA will not reveal the treatment codes until the end of the trial, when these data and the documents generated will be made available to the Principal Investigator (VA) and the Promoter (Institut d'investigació en Atenció Primària, IDIAP, Jordi Gol i Gurina ).

Statistical methods The description of the variables studied will be performed using conventional techniques. Variables with non-normal distribution will be transformed as necessary for normalization of distribution of values. The Kolmogorov-Smirnov and the Shapiro-Wilks test will be used to verify normality of distributions.

Analysis of the primary outcome The effects of iron dose supplement in each RCT on the biochemical iron status and mother-child health will be compared using regression models adjusted for those variables that can influence the relationship. Logistic regression or Cox models will be applied for qualitative variables such as, for example, the percentage of anemia or hemoconcentration at the end of pregnancy. Linear multiple regression models will be applied for dependent quantitative variables. The models will be adjusted for those variables that biologically affect the relationships studied, such as the serum ferritin levels, presence of alterations in the HFE gene, age of the mother, gestational age, parity, anthropometric indices, diet, and lifestyle, and the interactions between these variables. Initially included in the model will be all those variables that form part of the theoretical model and, in a second phase, the variables for entry into the model will be selected step by step (forward and backward) to achieve the most reduced stable models.

Conditions for the application of models will be verified using standard techniques that are based, essentially, on residuals analysis. The bilateral null hypothesis of normality, no difference, and non-significance of the regression coefficients, will be rejected when their

Monitoring To ensure correct conduct and security of the RCT according to the requirements of good clinical practice, external services will be contracted to perform the tasks of monitoring of the participating centers according to the requirements of the Spanish Agency of Medicines and Health Products [Agencia Española de Medicamentos y Productos Sanitarios; AEMPS].

ELIGIBILITY:
Inclusion Criteria:

* Adult woman
* ICS belonging to
* Pregnant less than 12 weeks gestation,
* To understand the Spanish or Catalan
* Sign the informed consent
* Without anemia (Hb <110 d / dL) in the pre-analytical at 12 weeks

Exclusion Criteria:

* Multiple or risk pregnancy.
* Taking iron supplements containing 10mg iron than in the previous three months
* Pregnant women with hypersensitivity to the active substance, hypersensitivity to egg proteins or intolerant to fructose or galactose.
* chronic or severe pre-existing disease that affects the nutritional development, such as cancer, diabetes mellitus and other metabolic diseases, malabsorptive diseases such as Crohn's disease, ulcerative colitis, gastro-duodenal ulcers, and liver diseases such as chronic hepatitis, liver cirrhosis and chronic pancreatitis.
* Immunosuppression: chronic HIV infection, transplant, neutropenic, or patients receiving immunosuppressive therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 704 (Actual)
Dates: Start 2013-07-10 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Anemia | at week 36 of gestation (3rd visit of study)
  - Anemia is defined as Hb <110 g/L in the 1st and 3rd trimester, Hb <110 in 2nd trimester (Centers for Disease Control and Prevention, 1998).
ferropenic anemia | at week 36 of gestation (3rd visit of study)
  - Ferropenic anemia is defined as: Hb < the normal limit, and serum ferritin (SF) <15 μg/L (WHO, 2007)
Risk of hemoconcentration | at week 36 of gestation (3rd visit of study)
  - Hemoconcentration risk is defined as: Hb >130 g/L in the 2nd and /or3rd trimester (Peña-Rosas y Viteri, 2009).

SECONDARY OUTCOMES:
C282Y polymorphisms of HFE gene | Blood analysis at 12 weeks of gestation.
  Presence or absence of polymorphisms: C282Y and H63D
Anthropometric parameters of newborn. | At birth
  weight (g)
Neurorconductual development of newborn (Bayley Scales) | 40days post-partum
  Units on a scale (score).
H63D polymorphisms of HFE gene | Blood analysis at 12 weeks of gestation.
  Presence or absence of polymorphisms: C282Y and H63D

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Arija, MD Professor, Study Director — Institut d'Investigació en Atenció Primària, IDIAP Jordi Gol i Gurina, Catalonia, Spain - Nutrition and Public Health Unit, Rovira i Virgili University
Locations (2):
- Spain (2):
  - Atención a la Salud Sexual y Reproductiva (ASSIR)- REUS- Altebrat, Reus, Tarragona
  - Atención a la Salud Sexual y Reproductiva (ASSIR)- Tarragona Valls, Tarragona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aranda N, Ribot B, Garcia E, Viteri FE, Arija V. Pre-pregnancy iron reserves, iron supplementation during pregnancy, and birth weight. Early Hum Dev. 2011 Dec;87(12):791-7. doi: 10.1016/j.earlhumdev.2011.06.003. Epub 2011 Jun 30. PMID 21723050
- [Background] Recommendations to prevent and control iron deficiency in the United States. Centers for Disease Control and Prevention. MMWR Recomm Rep. 1998 Apr 3;47(RR-3):1-29. PMID 9563847
- [Background] Hernandez-Martinez C, Canals J, Aranda N, Ribot B, Escribano J, Arija V. Effects of iron deficiency on neonatal behavior at different stages of pregnancy. Early Hum Dev. 2011 Mar;87(3):165-9. doi: 10.1016/j.earlhumdev.2010.12.006. Epub 2011 Jan 22. PMID 21256683
- [Background] Pena-Rosas JP, Viteri FE. Effects and safety of preventive oral iron or iron+folic acid supplementation for women during pregnancy. Cochrane Database Syst Rev. 2009 Oct 7;(4):CD004736. doi: 10.1002/14651858.CD004736.pub3. PMID 19821332
- [Background] Ribot B, Aranda N, Viteri F, Hernandez-Martinez C, Canals J, Arija V. Depleted iron stores without anaemia early in pregnancy carries increased risk of lower birthweight even when supplemented daily with moderate iron. Hum Reprod. 2012 May;27(5):1260-6. doi: 10.1093/humrep/des026. Epub 2012 Feb 21. PMID 22357769
- [Derived] Cendra-Duarte E, Canals J, Becerra-Tomas N, Mateu-Fabregat J, Bullo M, Arija V. Dietary glycemic index and load during pregnancy and offspring behavioral outcomes: exploring sex differences. Eur J Pediatr. 2025 Feb 6;184(2):178. doi: 10.1007/s00431-025-06005-y. PMID 39909936
- [Derived] Iglesias-Vazquez L, Gimeno M, Coronel P, Caspersen IH, Basora J, Arija V. Maternal factors associated with iron deficiency without anaemia in early pregnancy: ECLIPSES study. Ann Hematol. 2023 Apr;102(4):741-748. doi: 10.1007/s00277-023-05123-7. Epub 2023 Feb 15. PMID 36790457
- See also: World Health Organization (WHO). Iron and folate supplementation. Standards for maternal and neonatal care. Integrated Management of Pregnancy and Childbirth (IMPAC). Geneva: WHO, 2007; pp. 1-6. — http://whqlibdoc.who.int/hq/2007/a91272.pdf